CLINICAL TRIAL: NCT03945188
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, 52-Week Study to Assess the Efficacy and Safety of Etrasimod in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: Etrasimod Versus Placebo for the Treatment of Moderately to Severely Active Ulcerative Colitis
Acronym: ELEVATE UC 52
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD334-301; 2018-003985-15 (EudraCT Number)
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Results first posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-03

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Etrasimod; APD334
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etrasimod 2 mg (Experimental)
  Interventions: Drug: Etrasimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etrasimod — Etrasimod 2 mg tablet by mouth, once daily up to 52 weeks of treatment
  Other Names: APD334
  Arms: Etrasimod 2 mg
Drug: Placebo — Etrasimod matching placebo tablet by mouth, once daily up to 52 weeks of treatment
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether oral etrasimod is a safe and effective treatment for moderately to severely active ulcerative colitis.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosed with ulcerative colitis (UC) ≥ 3 months prior to screening
2. Active UC confirmed by endoscopy

Exclusion criteria:

1. Severe extensive colitis
2. Diagnosis of Crohn's disease (CD) or indeterminate colitis or the presence or history of a fistula consistent with CD
3. Diagnosis of microscopic colitis, ischemic colitis, or infectious colitis

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arena CT.gov Administrator, Study Director — Arena Pharmaceuticals
Locations (315):
- United States (67):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Arizona Digestive Health, Sun City, Arizona
  - Om Research, LLC, Lancaster, California
  - Entertainment Medical Group, Inc., Los Angeles, California
  - United Medical Doctors, Murrieta, California
  - San Diego Gastroenterology Medical Associates, San Diego, California
  - ACRC Studies, LLC, San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Gastro Florida, Clearwater, Florida
  - West Central Gastroenterology d/b/a Gastro Florida, Clearwater, Florida
  - Florida Center for Gastroenterology, Clearwater, Florida
  - Javier Sobrado, MD, Miami, Florida
  - Life Medical Center & Research, INC, Miami Lakes, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Office of Dr Meckstroth, Naples, Florida
  - NSB Research, New Smyrna Beach, Florida
  - Sarkis Clinical Trials - Parent, Ocala, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Theia Clinical Research, LLC, St. Petersburg, Florida
  - Advanced Research Institute, Inc., St. Petersburg, Florida
  - Lenus Research & Medical Group, Sweetwater, Florida
  - USF Physicians Group, Tampa, Florida
  - GCP Clinical Research, Tampa, Florida
  - Guardian Angel Research Center, Tampa, Florida
  - ASCLEPES Research Centers, P.C., Weeki Wachee, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Atlanta Gastroenterology Associates LLC, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Illinois Gastroenterology Group, Gurnee, Illinois
  - Gen1 Research, Moline, Illinois
  - Texas Digestive Disease Consultants, Baton Rouge, Louisiana
  - CroNOLA, Houma, Louisiana
  - Clinical Trials of SW Louisiana, LLC, Lake Charles, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Flint Clinical Research, Flint, Michigan
  - Robert Ferguson MD, West Bloomfield, Michigan
  - Gastrointestinal Associates, Flowood, Mississippi
  - Sierra Clinical Research, Las Vegas, Nevada
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Duke University Medical Center GI Clinical Research Unit, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Great Lakes Medical Research, LLC, Mentor, Ohio
  - Care Access Research, Poland, Ohio
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Great Lakes Medical Research, LLC, Harrisburg, Pennsylvania
  - GI for Kids, Knoxville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Coastal Medical Group, Baytown, Texas
  - Texas Gastroenterology Associates, PA, Cypress, Texas
  - Texas Digestive Disease Consultants, Dallas, Texas
  - Digestive Health Associates of Texas, Garland, Texas
  - CliniCore Texas, Houston, Texas
  - Baylor Gastroenterology Assoc, Houston, Texas
  - Biopharma Informatic, Inc. Research Center, Houston, Texas
  - Rio Grande Gastroenterology, McAllen, Texas
  - Biopharma Informatic, Inc. Research Center, Pasadena, Texas
  - Texas Digestive Disease Consultants - San Marcos, San Marcos, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Victoria Gastroenterology, Victoria, Texas
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Washington Gastroenterology, Bellevue, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Marshall University Department of Clinical Research, Huntington, West Virginia
  - Medical College of Wisconsin Clinical Trials Office, Milwaukee, Wisconsin
- Argentina (4):
  - Clinica Adventista Belgrano, CABA, Buenos Aires
  - Mautalen Salud e Investigacion, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Fundación Respirar- Centro Médico Dra. De Salvo, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - CICE Sanatorio 9 de Julio, San Miguel de Tucumán, Tucumán Province
- Australia (6):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Coastal Digestive Health Pty Ltd, Maroochydore, Queensland
  - Coral Sea Clinical Research Institute, North Mackay, Queensland
  - Austin Health Gastroenterology Department, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (3):
  - KH der Barmherzigen Brüder Linz, Linz
  - AKH - Medizinische Universität Wien, Vienna
  - Wilhelminenspital der Stadt Wien, Vienna
- Belarus (5):
  - Grodno City Clinical Hospital #4, Grodno
  - Institution "Gomel Regional Clinical Hospital", Homyel
  - Health Care Institution "10th City Clinical Hospital", Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
  - Vitebsk Regional Clinical Specialized Center, Vitebsk
- Belgium (4):
  - AZ Sint-Lucas & Volkskliniek, Ghent
  - UZ Gent Gastroenterology, Ghent
  - ZNA Jan Palfijn, Merksem
  - AZ Delta, Roeselare
- Bulgaria (11):
  - Medical center Medconsult Pleven OOD, Pleven
  - UMHAT Kanev AD, Ruse, Rousse
  - Diagnostic-Consultative Center I - Sliven, EOOD, Sliven
  - ACIBADEM CITY CLINIC TOKUDA HOSPITAL EAD,Clinical Research Center, Sofia
  - DCC "Alexandrovska", EOOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD,Clinic of gastroenterology, Sofia
  - UMHAT Tsaritsa Yoanna-ISUL EAD, Sofia
  - UMHATEM "N.I.Pirogov" EAD, Gastroenterology Department/Clinical Research center, next to the chimney, Sofia
  - Diagnostic Consultation Center CONVEX EOOD, Sofia
  - Acibadem City Clinic University Hospital EOOD, Sofia
  - Medical Center Nov Rehabilitatsionen Tsentar EOOD, Stara Zagora
- Mount Sinai Hospital, Toronto, Ontario, Canada
- Chile (5):
  - Enroll SpA, Santiago
  - Biomedica Research Group, Santiago
  - Hospital Sotero del Rio, Santiago
  - Centro de Investigación del Maule SPA, Talca
  - Clinical Research Chile SpA, Valdivia
- Croatia (7):
  - General Hospital "Dr.Tomislav Bardek" Koprivnica, Koprivnica
  - Clinical Hospital Centre Osijek, Osijek
  - General Hospital Zadar, Zadar
  - Clinical Hospital Dubrava, Zagreb
  - Clinical Hospital Sveti Duh, Zagreb
  - Polyclinic Bonifarm, Zagreb
  - University hospital centre Zagreb, Zagreb
- Czechia (8):
  - Fakultni nemocnice u svate Anny v Brne, Brno
  - Hepato-Gastroenterologie HK, s.r.o.,, Hradec Králové
  - GASTRO JeKa, s.r.o., Klatovy
  - PreventaMed s.r.o., Olomouc
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - ISCARE I.V.F. a.s., Prague
  - Nemocnice Na Bulovce, Prague
  - Nemocnice Slany, Slaný
- Denmark (2):
  - Aalborg University Hospital, department of medical gastroenterology, Aalborg, North Denmark
  - Herlev Hospital, Herlev
- Estonia (3):
  - Innomedica OÜ, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
- France (5):
  - CHU Nice - Hôpital de l'Archet 2, Nice, Alpes Maritimes
  - CHU Montpellier - HOPITAL SAINT-ELOI, Montpellier, Herault
  - CHU Nantes Hôtel-Dieu, Nantes, Loire Atlantique
  - CHU Grenoble Alpes - Hôpital Michallon, Grenoble
  - CHRU-Nancy Brabois, Vandœuvre-lès-Nancy
- Georgia (8):
  - LTD Acad. F. Todua Medical Center - LTD Research Institute of Clinical Medicine, Tbilisi
  - LTD Israeli-Georgian Medical Research clinic Helsicore, Tbilisi
  - LLC Vivamedi, Tbilisi
  - LTD Institute of Clinical Cardiology, Tbilisi
  - JSC Infectious Diseases, AIDS and Clinical Immunology Research Center, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LTD Central University Clinic After Academic N. Kipshidze, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center, Tbilisi
- Germany (7):
  - Praxis Dr. Joergensen, Remscheid, North Rhine-Westphalia
  - Schwerpunktpraxis Bonn, Bonn, Rhineland-Palatinate
  - Clinic for Internal Medicine I, University hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein
  - Krankenhaus Waldfriede, Berlin
  - Florence-Nightingale-Krankenhaus, Düsseldorf
  - Johanna Etienne Krankenhaus, Neuss
  - Klinische Forschung Schwerin GmbH, Schwerin
- Hungary (9):
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred
  - Bekes Megyei Kozpont Korhaz Dr Rethy Pal Tagkorhaz, 4. Belgyogyaszat es 2. Gasztroenterologia, Békéscsaba
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Bugat Pal Korhaz, Gyöngyös
  - SZTE AOK I.st dept. of Internal Medicine., Szeged
  - Clinfan Ltd. Outpatient Clinic, Szekszárd
  - 1th Dept of Gastroenterology, Szent Gyorgy Hospital, Székesfehérvár
  - Szent Borbala Korhaz, Tatabánya
- India (9):
  - Asian Institute of Gastroenterology, Hyderabad, Andhra Pradesh
  - Nirmal Hospitals Pvt Ltd, Surat, Gujarat
  - Surat Institute of Digestive Sciences, Surat, Gujarat
  - Fortis Memorial Research Institute, Gurgaon, Haryana
  - Aster Medcity,Aster DM healthcare Ltd, Kochi, Kerala
  - Midas Multispeciality Hospital-Nagpur, Nagpur, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Shweta Paliwal/Vipin Kumar Jain, Jaipur, Rajasthan
  - Postgraduate department of Medicine, GSVM Medical college, Kanpur, Uttar Pradesh
- Israel (9):
  - HaEmek Medical Center, Afula
  - Bnei Zion Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
- Italy (11):
  - Azienda Ospedaliera Saverio De Bellis, Castellana Grotte, Bari
  - Ospedale di Circolo, Rho, Milano
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese, Milano
  - Ospedale Sacro Cuore Don Calabria, Negrar, Verona
  - Spedali Civili di Brescia, U.O. Gastroenterologia, Brescia
  - Azienda Ospedaliera Ospedale Cannizzaro, Catania
  - Magna Graecia University, Catanzaro
  - A.O.U. Policlinico di Modena, Modena
  - Ospedale Sandro Pertini, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - CEMAD, Roma
  - Ospedale San Bortolo di Vicenza, Vicenza
- P. Stradins Clinical University Hospital, Riga, Latvia
- Saint George University Hospital Medical Center, Beirut, Lebanon
- Lithuania (5):
  - Kaunas Clinical Hospital, Kaunas
  - Klaipeda University Hospital, Department of Gastroenterology, Klaipėda
  - Republican Panevezys Hospital, Department of Gastroenterology, Panevezys
  - UAB "Inlita", Santaros Clinical Trials Centre, Vilnius
  - Vilnius University Hospital Santaros Clinics, Center of Hepatology, Gastroenterology and Dietology, Vilnius
- Mexico (5):
  - Centro de Investigacion Medico Biologica y Terapia Avanzada s.c., Guadalajara, Jalisco
  - InspirePharma S. de R. L. de C.V., Monterrey, Nuevo León
  - Scientia Investigación Clínica S.C., Chihuahua City
  - Hospital Angeles Chihuahua, Chihuahua City
  - Faicic S. de R.L. de Cv, Veracruz
- Moldova (4):
  - Clinical Hospital of the Ministry of Health, Labor and Social Protection, Chisinau
  - Rtl Sm Srl, Chisinau
  - Timofei Mosneaga Republican Clinical Hospital, Department of Gastroenterology, Chisinau
  - RTL SM SRL, Institutia Medico-Sanitara Publica Spitalul Clinic, Sectia Proctologie, Chisinau
- Netherlands (2):
  - Zuyderland Medisch Centrum - Sittard-Geleen, Geleen
  - ETZ Elisabeth, Tilburg
- Poland (21):
  - Centrum Dentystyczno-Lekarskie Promedica Joanna Markiewicz, Będzin
  - Gastromed Kralisz, Romatowski, Stachurska sp.j, Bialystok
  - Centrum Medyczne Pratia Czestochowa, Częstochowa
  - Karkonoskie Centrum Badan Klinicznych Lexmedica, Jelenia Góra
  - Topolowa Medicenter Mrozek & Wspolnicy Spolka Jawna, Krakow
  - AmiCare Sp. z O.O. Sp.K., Lodz
  - IP Clinic, Lodz
  - Med-Gastr Przychodnia Specjalistyczna, Lodz
  - Allmedica Badania Kliniczne Sp. z o.o. Sp.k., Nowy Targ
  - Medicenter Nowy Targ, Nowy Targ
  - Medicome Sp. Zo.O., Oświęcim
  - Centrum Medyczne Grunwald, Poznan
  - SOLUMED Centrum Medyczne, Poznan
  - Centrum Medyczne Medyk, Rzeszów
  - ENDOSKOPIA Sp.zo.o, Sopot
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
  - EMC INSTYTUT MEDYCZNY SA, EuroMediCare Szpital Specjalistyczny z Przychodnia - Dzial Farmacji, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - Jerzy Rozciecha- Lexmedica, Wroclaw
- Portugal (4):
  - Hospital de Braga, Braga
  - Centro Hospitalar e Universitário de Coimbra Serviço Gastrenterologia, Coimbra
  - Centro Hospitalar de São João, EPE, Porto
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E., Vila Nova de Gaia
- Romania (12):
  - S.C Policlinica CCBR S.R.L, Bucharest
  - S.C MedLife SA, Bucharest
  - Dr. Carol Davila Central University Emergency Military Hospital, Bucharest
  - Delta Health Care srl, Bucharest
  - S.C Euroclinic Hospital S.A, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Centrul Medical Unirea srl, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta, Craiova
  - Cabinet Medical Dr. Fratila S.R.L, Oradea
  - S.C Pelican Impex S.R.L, Oradea
- Russia (19):
  - LLC "Multidisciplinary Medical Clinic "Anthurium", Barnaul
  - LLC "Alyans Biomedical- Ural Group", Irkutsk
  - Kazan State Medical University, Kazan'
  - SAIH "Kemerovo Regional Clinical Hospital, Kemerovo
  - SBIH of Nizhniy Novgorod region "Nizhniy Novgorod Regional Clinical Hospital n.a. N.A. Semashko", Nizhny Novgorod
  - LLC Medicine Center SibNovoMed, Novosibirsk
  - CDC Ultramed, Omsk
  - State Budgetary Healthcare Institution "Penza Region Clinical Hospital n.a. N.N. Burdenko", Penza
  - LLC "Medinet", Saint Petersburg
  - Federal state Budgetary Educational Institution of Higher Education "North-Western Medical University", Saint Petersburg
  - LLC SM-Clinic, Saint Petersburg
  - LLC "Gastroenterological centre Expert", Saint Petersburg
  - Irkutsk State Medical Academy of Continuing Education, Samara
  - Private Educational Institution of Higher Education "Medical University REAVIZ", Samara
  - LLC Medical Company "Hepatologist", Samara
  - SPb SBIH "City Hospital # 40 of Kurortnyi region", Sestroretsk
  - LLC Uromed, Smolensk
  - Stavropol Regional Clinical Diagnostic Centre, Stavropol
  - LLC "Polyclinic of ultrasonography 4D", Stavropol
- Serbia (5):
  - Clinical Center " Dr Dragisa Misovic Dedinje", Belgrade
  - Clinical Center of Serbia, Belgrade
  - Clinical Health Center Zvezdara, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - General Hospital Sremska Mitrovica, Sremska Mitrovica
- Slovakia (8):
  - ENDOMED, s.r.o., Vranov nad Topľou, Presov
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica, Banská Bystrica
  - Alian S.R.O, Bardejov
  - KM Management spol. s r.o., Nitra
  - Fakultna nemocnica Nitra, Nitra
  - GASTROENTEROLOG, s.r.o., Nové Zámky
  - Gastro I, s.r.o., Prešov
  - Accout Center s.r.o., Šahy
- South Africa (4):
  - Johese Clinical Research: Unitas, Lyttelton, Centurion
  - Johese Clinical Research, Midstream, Centurion
  - Lenasia Clinical Trial Centre, Johannesburg, Gauteng
  - Dr JP Wright Practice, Cape Town, Western Cape
- South Korea (6):
  - Kyungpook National University Hospital, Junggu, Daegu
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul, Seodaemun-gu
  - Dong-A University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
- Hospital Universitario La Paz, Madrid, Spain
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- Thailand (4):
  - Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok
  - Supaporn Lertkawinanan, Pathum Wan, Bangkok
  - Phramongkutklao Hospital, Ratchathewi, Bangkok
  - Ms. Arawan Larplertsakul, Chiang Mai
- Turkey (Türkiye) (4):
  - Uludag University Medical Faculty, Beşevler, Yenimahalle / Ankara
  - Gazi University Medical Faculty, Ankara
  - Antalya Training and Research Hospital, Antalya
  - Kocaeli University Research and Training Hospital, Kocaeli
- Ukraine (17):
  - I.I.Mechnykov Dnipropetrovsk Regional Clinical Hospital, Dnipro
  - Department of Propaedeutics of Internal Medicine Ivano-Frankivsk National Medical University, Ivano-Frankivsk
  - Municipal non-profit enterprise "Regional Clinical Hospital of Ivano-Frankivsk Regional Council", Ga, Ivano-Frankivsk
  - CNE Prof. O.O. Shalimov Kharkiv City Clinical Hospital #2 of KCC, Kharkiv
  - Communal Non-commercial Enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - Communal Non-Commercial Enterprise City Clinical Hospital #13 of Kharkiv City Council, Kharkiv
  - Communal Noncommercial Enterprise Ye.Ye. Karabelesh Kherson City Clinical Hospital of Kherson City, Kherson
  - Kremenchuk first city hospital n.a. O.T. Bohaievskyi, Kremenchuk
  - National Military Medical Clinical Center Main Military Clinical Hospital, Kyiv
  - Kyiv City Clinical Hospital N 1, Kyiv
  - Communal Non-Commercial Enterprise Lviv Clinical Hospital of Emergency Medical Care, Lviv
  - Odesa regional clinical hospital, regional center of gastroenterology, surgical department, Odesa
  - A. Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - Medical Clinical Investigational Center of Medical Center Health Clinic LLC, Vinnytsia
  - M.I. Pyrogov VRCH Dept of Gastroenterology M.I. Pyrogov VNMU, Vinnytsia
  - SRI of Invalid Rehabilitation (EST Complex) of Vinnytsia M.I.Pyrogov NMU MOHU, Vinnytsia
  - Communal Institution City Clinical Hospital #6, Department of Gastroenterology, Zaporizhzhia
- United Kingdom (6):
  - Barts Health NHS Trust - Whipps Cross University Hospital, London, Greater London
  - Guys and St Thomas NHS Foundation Trust, London, Greater London
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk
  - Yeovil Hospital NHS Foundation Trust, Yeovil, Somerset
  - Belfast Health and Social Care Trust Royal Victoria Hospital, Belfast
  - West Hertfordshire Hospitals NHS Trust Hemel Hempstead General Hospital, Hemel Hempstead

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dubinsky MC, Chaparro M, Irving PM, Hur P, Sidhu S, Woolcott JC, Wang W, Goetsch M, Torres J, Panaccione R. Rapid symptomatic improvement with etrasimod in ulcerative colitis: a post-hoc analysis of the ELEVATE UC program. Inflamm Bowel Dis. 2026 Feb 8:izaf333. doi: 10.1093/ibd/izaf333. Online ahead of print. PMID 41655066
- [Derived] Chaparro M, Panaccione R, Sands BE, Irving PM, Goetsch M, Kunina E, Wang W, Wu J, Woolcott JC, Bartolome L, Cognata C, Wosik K, Dubinsky MC. Etrasimod for the symptomatic relief of ulcerative colitis: a post-hoc analysis from the ELEVATE UC clinical programme. BMJ Open Gastroenterol. 2025 Aug 31;12(1):e001838. doi: 10.1136/bmjgast-2025-001838. PMID 40889900
- [Derived] Yarur AJ, Reinisch W, Chang S, Gecse KB, Green J, Abbatemarco AM, Wu J, Goetsch M, Lazin K, Pradeep G, Sands BE. Efficacy of Etrasimod in Ulcerative Colitis: Analysis of ELEVATE UC 52 and ELEVATE UC 12 by Baseline Endoscopic Severity. Clin Gastroenterol Hepatol. 2026 Jan;24(1):210-220.e3. doi: 10.1016/j.cgh.2025.06.020. Epub 2025 Jul 4. PMID 40618942
- [Derived] Lichtenstein GR, Allegretti JR, Loftus EV Jr, Irving PM, Banerjee R, Charabaty A, Kuehbacher T, Bananis E, Woolcott JC, Dalam AB, Lazin K, Keating M, McDonnell A, Danese S. Assessment and Impact of Age on the Safety and Efficacy of Etrasimod in Patients With Ulcerative Colitis: A Post Hoc Analysis of Data From the ELEVATE UC Clinical Program. Inflamm Bowel Dis. 2025 Sep 1;31(9):2352-2362. doi: 10.1093/ibd/izae308. PMID 40184206
- [Derived] Sands BE, Dubinsky MC, Kotze PG, Vermeire S, Panaccione R, Long MD, Woolcott JC, Wu J, McDonnell A, Goetsch M, Bananis E, Yarur AJ. Efficacy and Safety of Etrasimod in Patients With Moderately to Severely Active Ulcerative Colitis Stratified by Baseline Modified Mayo Score: A Post Hoc Analysis From the Phase 3 ELEVATE UC Clinical Program. Inflamm Bowel Dis. 2025 Oct 1;31(10):2681-2692. doi: 10.1093/ibd/izaf036. PMID 40036804
- [Derived] Afzali A, Regueiro M, Yarur AJ, Zabana Y, Ng SC, Menon S, McDonnell A, Lazin K, Keating M, Bhattacharjee A, Branquinho D, Bananis E, Peyrin-Biroulet L. Concomitant Use of Etrasimod With Opioids or Antidepressants in Patients With Ulcerative Colitis-A Safety Analysis. United European Gastroenterol J. 2025 Jun;13(5):719-727. doi: 10.1002/ueg2.12745. Epub 2025 Feb 1. PMID 39891572
- [Derived] Yarur AJ, Long MD, Torres J, Nandi N, Cross RK, Abbatemarco AM, Blanco D, Niezychowski W, Crosby C, Wu J, Pradeep G, Goetsch M, Panaccione R. Body Mass Index Did Not Affect Efficacy and Safety of Etrasimod: A Post Hoc Analysis of the ELEVATE Ulcerative Colitis Clinical Program. Am J Gastroenterol. 2025 Nov 1;120(11):2611-2622. doi: 10.14309/ajg.0000000000003330. Epub 2025 Jan 29. PMID 39878434
- [Derived] Vermeire S, Rubin DT, Peyrin-Biroulet L, Dubinsky MC, Regueiro M, Irving PM, Goetsch M, Lazin K, Gu G, Wu J, Modesto I, McDonnell A, Guo X, Green J, Dalam AB, Yarur AJ. Cardiovascular events observed among patients in the etrasimod clinical programme: an integrated safety analysis of patients with moderately to severely active ulcerative colitis. BMJ Open Gastroenterol. 2025 Jan 8;12(1):e001516. doi: 10.1136/bmjgast-2024-001516. PMID 39778975
- [Derived] Yarur AJ, Chiorean MV, Allegretti JR, Cross RK, Ha C, Goetsch M, McDonnell A, Dalam AB, Wu J, Blanco DA, Abbatemarco AM, Panes J. Etrasimod as a Monotherapy or With Concomitant Use of Corticosteroids and/or Aminosalicylates: Results From the ELEVATE UC Clinical Program. Inflamm Bowel Dis. 2025 Aug 1;31(8):2144-2153. doi: 10.1093/ibd/izae288. PMID 39671695
- [Derived] Lees CW, Torres J, Leung Y, Vermeire S, Fellmann M, Modesto I, McDonnell A, Lazin K, Keating M, Goetsch M, Wu J, Loftus EV Jr. Non-serious adverse events in patients with ulcerative colitis receiving etrasimod: an analysis of the phase II OASIS and phase III ELEVATE UC 52 and ELEVATE UC 12 clinical trials. Therap Adv Gastroenterol. 2024 Nov 7;17:17562848241293643. doi: 10.1177/17562848241293643. eCollection 2024. PMID 39526078
- [Derived] Armuzzi A, Rubin DT, Schreiber S, Panes J, Fellmann M, Bartolome L, Gruben D, Goetsch M, Bhattacharjee A, Chaparro M, Dubinsky MC. Health-Related Quality of Life Outcomes With Etrasimod Treatment in Patients With Ulcerative Colitis: A Post Hoc Analysis of Data From ELEVATE UC 52 and ELEVATE UC 12. Inflamm Bowel Dis. 2025 Jun 13;31(6):1583-1594. doi: 10.1093/ibd/izae229. PMID 39326009
- [Derived] Sands BE, Leung Y, Rubin DT, Gecse KB, Panes J, Goetsch M, Wang W, Woolcott JC, Smith CC, Wosik K, Schreiber S. Etrasimod Corticosteroid-Free Efficacy, Impact of Concomitant Corticosteroids on Efficacy and Safety, and Corticosteroid-Sparing Effect in Ulcerative Colitis: Analyses of the ELEVATE UC Clinical Program. J Crohns Colitis. 2025 Mar 5;19(3):jjae150. doi: 10.1093/ecco-jcc/jjae150. PMID 39306680
- [Derived] Magro F, Peyrin-Biroulet L, Sands BE, Danese S, Jairath V, Goetsch M, Bhattacharjee A, Wu J, Branquinho D, Modesto I, Feagan BG. Endoscopic, Histologic, and Composite Endpoints in Patients With Ulcerative Colitis Treated With Etrasimod. Clin Gastroenterol Hepatol. 2025 Feb;23(2):341-350.e6. doi: 10.1016/j.cgh.2024.07.010. Epub 2024 Jul 31. PMID 39089519
- [Derived] Vermeire S, Sands BE, Peyrin-Biroulet L, D'Haens GR, Panes J, Yarur AJ, Wolf DC, Ritter T, Schreiber S, Woolcott JC, Modesto I, Keating M, Shan K, Wu J, Chiorean MV, Baert F, Dubinsky MC, Goetsch M, Danese S, Feagan BG. Impact of Prior Biologic or Janus Kinase Inhibitor Therapy on Efficacy and Safety of Etrasimod in the ELEVATE UC 52 and ELEVATE UC 12 Trials. J Crohns Colitis. 2024 Nov 4;18(11):1780-1794. doi: 10.1093/ecco-jcc/jjae079. PMID 38877972
- [Derived] Regueiro M, Siegmund B, Yarur AJ, Steinwurz F, Gecse KB, Goetsch M, Bhattacharjee A, Wu J, Green J, McDonnell A, Crosby C, Lazin K, Branquinho D, Modesto I, Abreu MT. Etrasimod for the Treatment of Ulcerative Colitis: Analysis of Infection Events from the ELEVATE UC Clinical Programme. J Crohns Colitis. 2024 Oct 15;18(10):1596-1605. doi: 10.1093/ecco-jcc/jjae060. PMID 38700040
- [Derived] Peyrin-Biroulet L, Dubinsky MC, Sands BE, Panes J, Schreiber S, Reinisch W, Feagan BG, Danese S, Yarur AJ, D'Haens GR, Goetsch M, Wosik K, Keating M, Lazin K, Wu J, Modesto I, McDonnell A, Bartolome L, Vermeire S. Efficacy and Safety of Etrasimod in Patients with Moderately to Severely Active Isolated Proctitis: Results From the Phase 3 ELEVATE UC Clinical Programme. J Crohns Colitis. 2024 Aug 14;18(8):1270-1282. doi: 10.1093/ecco-jcc/jjae038. PMID 38613425
- [Derived] Sandborn WJ, Vermeire S, Peyrin-Biroulet L, Dubinsky MC, Panes J, Yarur A, Ritter T, Baert F, Schreiber S, Sloan S, Cataldi F, Shan K, Rabbat CJ, Chiorean M, Wolf DC, Sands BE, D'Haens G, Danese S, Goetsch M, Feagan BG. Etrasimod as induction and maintenance therapy for ulcerative colitis (ELEVATE): two randomised, double-blind, placebo-controlled, phase 3 studies. Lancet. 2023 Apr 8;401(10383):1159-1171. doi: 10.1016/S0140-6736(23)00061-2. Epub 2023 Mar 2. PMID 36871574

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderately to severely active ulcerative colitis (UC) were enrolled in this study. Eligible participants were randomized in a 2:1 ratio to receive either etrasimod 2 milligrams (mg) once daily or matching placebo once daily for up to 52 weeks.
Pre-assignment Details: The study included a Screening Period (up to 28 days), a 12-Week Treatment Period (induction) followed by a 40-Week Treatment Period (maintenance; for which no re-randomization took place), and a 2-Week and 4-Week Follow-Up Period.
Groups:
- Etrasimod 2 mg: Etrasimod 2 mg was administered orally once daily for up to 52 weeks.
- Placebo: Placebo was administered orally once daily for up to 52 weeks.
Period: Overall Study
Arm/Group | Etrasimod 2 mg | Placebo
Started | 289 | 144
Completed | 161 | 46
Not Completed | 128 | 98
Not completed — Protocol Violation | 1 | 0
Not completed — Disease worsening | 79 | 73
Not completed — Physician Decision | 2 | 2
Not completed — Lack of Efficacy | 7 | 4
Not completed — Pregnancy | 2 | 0
Not completed — Withdrawal by participant or parent/guardian | 24 | 10
Not completed — Adverse Event | 10 | 5
Not completed — Other | 2 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Etrasimod 2 mg | Placebo | Total
Number analyzed (Participants) | 289 | 144 | 433
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 272 | 133 | 405
  >=65 years | 17 | 10 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (13.97) | 38.9 (14.04) | 40.4 (14.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 56 | 193
  Male | 152 | 88 | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 275 | 136 | 411
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 22 | 9 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 256 | 129 | 385
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Remission at Week 12
Description: Clinical remission was based on the modified Mayo score (MMS). The MMS is a composite score of 3 assessments consisting of participant-reported symptoms using daily eDiary and centrally read endoscopy: stool frequency (SF), rectal bleeding (RB) and endoscopic score (ES). Clinical remission was defined as SF subscore = 0 (or = 1 with a ≥ 1-point decrease from Baseline), RB subscore = 0, and ES ≤ 1 (excluding friability). Each component subscore ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: At Week 12
Population: FAS (consisting of all randomized participants who received at least 1 dose of study treatment) with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 27.0 | 7.4
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 19.75, 95% CI 2-sided [12.88 to 26.63]

2. Primary Outcome: Percentage of Participants Achieving Clinical Remission at Week 52
Description: Clinical remission was based on the MMS which is a composite score of 3 assessments: SF, RB and ES. Clinical remission was defined as SF subscore = 0 (or = 1 with a ≥ 1-point decrease from Baseline), RB subscore = 0, and ES ≤ 1 (excluding friability). Each component subscore ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: At Week 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 32.1 | 6.7
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 25.39, 95% CI 2-sided [18.42 to 32.36]

3. Secondary Outcome: Percentage of Participants Achieving Endoscopic Improvement at Week 12
Description: Endoscopic improvement was defined as an ES ≤ 1 (excluding friability). The ES ranged from 0 to 3 (where 0 = normal/inactive disease and 3 = severe disease).
Time Frame: At Week 12
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 35.0 | 14.1
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 21.18, 95% CI 2-sided [13.03 to 29.32]

4. Secondary Outcome: Percentage of Participants Achieving Endoscopic Improvement at Week 52
Description: as for outcome 3
Time Frame: At Week 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 37.2 | 10.4
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 26.69, 95% CI 2-sided [18.99 to 34.39]

5. Secondary Outcome: Percentage of Participants Achieving Symptomatic Remission at Week 12
Description: Symptomatic remission was defined as an SF subscore = 0 (or = 1 with a ≥ 1-point decrease from Baseline) and RB subscore = 0. The SF subscore ranged from 0 to 3 (where 0 = normal number of stools and 3 = at least 5 stools more than normal) and RB subscore ranged from 0 to 3 (where 0 = no blood and 3 = blood alone passes). Higher scores indicate more severe disease.
Time Frame: At Week 12
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 46.0 | 21.5
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 24.55, 95% CI 2-sided [15.46 to 33.63]

6. Secondary Outcome: Percentage of Participants Achieving Symptomatic Remission at Week 52
Description: as for outcome 5
Time Frame: At Week 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 43.4 | 18.5
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 24.89, 95% CI 2-sided [16.17 to 33.60]

7. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 12
Description: Mucosal healing was defined as an ES ≤ 1 (excluding friability) with histologic remission measured by a Geboes Index score < 2.0. The ES ranged from 0 to 3 (where 0 = normal/inactive disease and 3 = severe disease). The Geboes score grading system is a validated score for evaluating histologic disease activity in UC as follows: grade 0 = structural and architectural changes; grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher Geboes score indicates more severe disease.
Time Frame: At Week 12
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 21.2 | 4.4
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.88, 95% CI 2-sided [10.78 to 22.98]

8. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 52
Description: as for outcome 7
Time Frame: At Week 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 26.6 | 8.1
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 18.39, 95% CI 2-sided [11.39 to 25.39]

9. Secondary Outcome: Percentage of Participants Achieving Corticosteroid-free Clinical Remission at Week 52
Description: Corticosteroid-free clinical remission was defined as an SF subscore = 0 (or = 1 with a ≥ 1-point decrease from Baseline), RB subscore = 0, ES ≤ 1 (excluding friability), and have not received corticosteroids for ≥ 12 weeks in the 40-Week Treatment Period. Each component subscore ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: At Week 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 32.1 | 6.7
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 25.39, 95% CI 2-sided [18.42 to 32.36]

10. Secondary Outcome: Percentage of Participants Achieving Sustained Clinical Remission at Both Weeks 12 and 52
Description: Sustained clinical remission was defined as an SF subscore = 0 (or = 1 with a ≥ 1-point decrease from Baseline), RB subscore = 0, and ES ≤ 1 (excluding friability) at both Week 12 and Week 52. Each component subscore ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: At Weeks 12 and 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 17.9 | 2.2
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.84, 95% CI 2-sided [10.66 to 21.03]

11. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 12
Description: Clinical response was based on the MMS which is a composite score of 3 assessments: SF, RB and ES. Clinical response was defined as a ≥ 2-point and ≥ 30% decrease from Baseline MMS, and a ≥ 1-point decrease from Baseline in RB subscore or an absolute RB subscore ≤ 1. Each component subscore ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: At Week 12
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 62.4 | 34.1
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 28.27, 95% CI 2-sided [18.51 to 38.02]

12. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 52
Description: Clinical response was based on the MMS which is a composite score of 3 assessments: SF, RB and ES. Clinical response was defined as a ≥ 2-point and ≥ 30% decrease from Baseline MMS, and a ≥ 1-point decrease from Baseline in RB subscore or an absolute RB sub-score ≤ 1. Each component subscore ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: At Week 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 48.2 | 23.0
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 24.93, 95% CI 2-sided [15.79 to 34.07]

13. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Both Weeks 12 and 52
Description: as for outcome 11
Time Frame: At Weeks 12 and 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 44.9 | 18.5
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 26.16, 95% CI 2-sided [17.48 to 34.84]

14. Secondary Outcome: Percentage of Participants With Mucosal Healing at Both Weeks 12 and 52
Description: as for outcome 7
Time Frame: At Weeks 12 and 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 13.5 | 2.2
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 11.32, 95% CI 2-sided [6.49 to 16.14]

15. Secondary Outcome: Percentage of Participants Achieving Endoscopic Normalization at Week 12
Description: Endoscopic normalization was defined as an ES = 0. The ES ranged from 0 to 3 (where 0= normal/inactive disease and 3= severe disease).
Time Frame: At Week 12
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 14.6 | 4.4
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.23, 95% CI 2-sided [4.73 to 15.73]

16. Secondary Outcome: Percentage of Participants Achieving Endoscopic Normalization at Week 52
Description: as for outcome 15
Time Frame: At Week 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 26.3 | 5.9
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.39, 95% CI 2-sided [13.79 to 26.98]

17. Secondary Outcome: Percentage of Participants Achieving Endoscopic Normalization at Both Weeks 12 and 52
Description: as for outcome 15
Time Frame: At Weeks 12 and 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants | 10.6 | 1.5
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 9.16, 95% CI 2-sided [4.93 to 13.38]

18. Secondary Outcome: Percentage of Participants Achieving Symptomatic Remission by Study Visit
Description: as for outcome 5
Time Frame: At Weeks 2, 4, 8, 16, 20, 24, 32, 40, and 48
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants
  Week 2 | 15.3 | 8.9
  Week 4 | 28.1 | 13.3
  Week 8 | 37.6 | 20.7
  Week 16 | 43.1 | 21.5
  Week 20 | 43.8 | 20.0
  Week 24 | 44.9 | 23.7
  Week 32 | 44.5 | 18.5
  Week 40 | 42.0 | 18.5
  Week 48 | 42.0 | 15.6
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 2; Test type: Superiority; p = 0.049, Cochran-Mantel-Haenszel; Risk Difference (RD) = 6.49, 95% CI 2-sided [0.02 to 12.95]
Statistical Analysis 2: Comparison: Etrasimod 2 mg vs Placebo; Week 4; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.03, 95% CI 2-sided [7.32 to 22.74]
Statistical Analysis 3: Comparison: Etrasimod 2 mg vs Placebo; Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.85, 95% CI 2-sided [8.06 to 25.63]
Statistical Analysis 4: Comparison: Etrasimod 2 mg vs Placebo; Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 21.66, 95% CI 2-sided [12.71 to 30.61]
Statistical Analysis 5: Comparison: Etrasimod 2 mg vs Placebo; Week 20; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 23.74, 95% CI 2-sided [14.98 to 32.51]
Statistical Analysis 6: Comparison: Etrasimod 2 mg vs Placebo; Week 24; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 21.04, 95% CI 2-sided [11.83 to 30.24]
Statistical Analysis 7: Comparison: Etrasimod 2 mg vs Placebo; Week 32; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 25.82, 95% CI 2-sided [17.08 to 34.56]
Statistical Analysis 8: Comparison: Etrasimod 2 mg vs Placebo; Week 40; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 23.47, 95% CI 2-sided [14.80 to 32.14]
Statistical Analysis 9: Comparison: Etrasimod 2 mg vs Placebo; Week 48; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 26.37, 95% CI 2-sided [17.92 to 34.82]

19. Secondary Outcome: Percentage of Participants Achieving Complete Symptomatic Remission by Study Visit
Description: Complete symptomatic remission was defined as an SF subscore = 0 and RB subscore = 0. The SF subscore ranged from 0 to 3 (where 0 = normal number of stools and 3 = at least 5 stools more than normal) and RB subscore ranged from 0 to 3 (where 0 = no blood and 3 = blood alone passes). Higher scores indicate more severe disease.
Time Frame: At Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48 and 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants
  Week 2 | 5.8 | 2.2
  Week 4 | 11.3 | 4.4
  Week 8 | 16.8 | 6.7
  Week 12 | 23.0 | 6.7
  Week 16 | 21.2 | 5.9
  Week 20 | 22.3 | 4.4
  Week 24 | 22.3 | 8.1
  Week 32 | 23.0 | 3.0
  Week 40 | 21.2 | 5.9
  Week 48 | 19.7 | 2.2
  Week 52 | 24.5 | 4.4
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 2; Test type: Superiority; p = 0.057, Cochran-Mantel-Haenszel; Risk Difference (RD) = 3.59, 95% CI 2-sided [-0.11 to 7.30]
Statistical Analysis 2: Comparison: Etrasimod 2 mg vs Placebo; Week 4; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Risk Difference (RD) = 6.88, 95% CI 2-sided [1.86 to 11.90]
Statistical Analysis 3: Comparison: Etrasimod 2 mg vs Placebo; Week 8; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.14, 95% CI 2-sided [4.09 to 16.20]
Statistical Analysis 4: Comparison: Etrasimod 2 mg vs Placebo; Week 12; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 16.36, 95% CI 2-sided [9.89 to 22.83]
Statistical Analysis 5: Comparison: Etrasimod 2 mg vs Placebo; Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.37, 95% CI 2-sided [9.23 to 21.52]
Statistical Analysis 6: Comparison: Etrasimod 2 mg vs Placebo; Week 20; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.80, 95% CI 2-sided [11.85 to 23.75]
Statistical Analysis 7: Comparison: Etrasimod 2 mg vs Placebo; Week 24; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 14.24, 95% CI 2-sided [7.45 to 21.04]
Statistical Analysis 8: Comparison: Etrasimod 2 mg vs Placebo; Week 32; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.03, 95% CI 2-sided [14.25 to 25.81]
Statistical Analysis 9: Comparison: Etrasimod 2 mg vs Placebo; Week 40; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 15.13, 95% CI 2-sided [8.91 to 21.35]
Statistical Analysis 10: Comparison: Etrasimod 2 mg vs Placebo; Week 48; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.52, 95% CI 2-sided [12.16 to 22.87]
Statistical Analysis 11: Comparison: Etrasimod 2 mg vs Placebo; Week 52; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 19.86, 95% CI 2-sided [13.75 to 25.98]

20. Secondary Outcome: Percentage of Participants Achieving Non-invasive Clinical Response by Study Visit
Description: Non-invasive clinical response was defined as a ≥ 30% decrease from Baseline in composite RB and SF subscores, and a ≥ 1-point decrease from Baseline in RB subscore or RB subscore ≤ 1. The SF subscore ranged from 0 to 3 (where 0 = normal number of stools and 3 = at least 5 stools more than normal) and RB subscore ranged from 0 to 3 (where 0 = no blood and 3 = blood alone passes). The composite RB and SF score range was from 0 to 6, with higher scores indicating more severe disease.
Time Frame: At Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants
  Week 2 | 38.3 | 33.3
  Week 4 | 56.2 | 39.3
  Week 8 | 63.1 | 43.0
  Week 12 | 65.7 | 42.2
  Week 16 | 55.5 | 30.4
  Week 20 | 57.3 | 28.1
  Week 24 | 56.6 | 30.4
  Week 32 | 54.0 | 25.2
  Week 40 | 51.5 | 23.0
  Week 48 | 51.1 | 21.5
  Week 52 | 50.4 | 23.7
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 2; Test type: Superiority; p = 0.336, Cochran-Mantel-Haenszel; Risk Difference (RD) = 4.83, 95% CI 2-sided [-5.01 to 14.68]
Statistical Analysis 2: Comparison: Etrasimod 2 mg vs Placebo; Week 4; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.11, 95% CI 2-sided [7.06 to 27.15]
Statistical Analysis 3: Comparison: Etrasimod 2 mg vs Placebo; Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.17, 95% CI 2-sided [10.15 to 30.19]
Statistical Analysis 4: Comparison: Etrasimod 2 mg vs Placebo; Week 12; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 23.44, 95% CI 2-sided [13.45 to 33.43]
Statistical Analysis 5: Comparison: Etrasimod 2 mg vs Placebo; Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 25.25, 95% CI 2-sided [15.67 to 34.83]
Statistical Analysis 6: Comparison: Etrasimod 2 mg vs Placebo; Week 20; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 29.20, 95% CI 2-sided [19.77 to 38.64]
Statistical Analysis 7: Comparison: Etrasimod 2 mg vs Placebo; Week 24; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 26.08, 95% CI 2-sided [16.47 to 35.69]
Statistical Analysis 8: Comparison: Etrasimod 2 mg vs Placebo; Week 32; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 28.68, 95% CI 2-sided [19.35 to 38.02]
Statistical Analysis 9: Comparison: Etrasimod 2 mg vs Placebo; Week 40; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 28.43, 95% CI 2-sided [19.30 to 37.55]
Statistical Analysis 10: Comparison: Etrasimod 2 mg vs Placebo; Week 48; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 29.59, 95% CI 2-sided [20.55 to 38.64]
Statistical Analysis 11: Comparison: Etrasimod 2 mg vs Placebo; Week 52; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 26.43, 95% CI 2-sided [17.18 to 35.68]

21. Secondary Outcome: Percentage of Participants Achieving Symptomatic Response by Study Visit
Description: Symptomatic response was defined as a ≥ 30% decrease from Baseline in composite RB and SF subscores. The SF subscore ranged from 0 to 3 (where 0= normal number of stools and 3= at least 5 stools more than normal) and RB subscore ranged from 0 to 3 (where 0= no blood and 3= blood alone passes). The composite RB and SF score range was from 0 to 6, with higher scores indicating more severe disease.
Time Frame: At Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: FAS with actual Baseline MMS 5 to 9.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 274 | 135
Percentage of participants
  Week 2 | 39.4 | 33.3
  Week 4 | 57.3 | 40.0
  Week 8 | 64.6 | 43.7
  Week 12 | 66.4 | 42.2
  Week 16 | 55.5 | 31.1
  Week 20 | 57.7 | 28.1
  Week 24 | 56.9 | 30.4
  Week 32 | 54.7 | 25.2
  Week 40 | 51.8 | 23.0
  Week 48 | 51.5 | 21.5
  Week 52 | 50.7 | 23.7
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Week 2; Test type: Superiority; p = 0.240, Cochran-Mantel-Haenszel; Risk Difference (RD) = 5.93, 95% CI 2-sided [-3.96 to 15.81]
Statistical Analysis 2: Comparison: Etrasimod 2 mg vs Placebo; Week 4; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 17.50, 95% CI 2-sided [7.48 to 27.53]
Statistical Analysis 3: Comparison: Etrasimod 2 mg vs Placebo; Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.93, 95% CI 2-sided [10.92 to 30.94]
Statistical Analysis 4: Comparison: Etrasimod 2 mg vs Placebo; Week 12; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 24.13, 95% CI 2-sided [14.15 to 34.10]
Statistical Analysis 5: Comparison: Etrasimod 2 mg vs Placebo; Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 24.51, 95% CI 2-sided [14.89 to 34.13]
Statistical Analysis 6: Comparison: Etrasimod 2 mg vs Placebo; Week 20; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 29.57, 95% CI 2-sided [20.13 to 39.01]
Statistical Analysis 7: Comparison: Etrasimod 2 mg vs Placebo; Week 24; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 26.45, 95% CI 2-sided [16.88 to 36.02]
Statistical Analysis 8: Comparison: Etrasimod 2 mg vs Placebo; Week 32; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 29.35, 95% CI 2-sided [20.01 to 38.68]
Statistical Analysis 9: Comparison: Etrasimod 2 mg vs Placebo; Week 40; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 28.83, 95% CI 2-sided [19.71 to 37.95]
Statistical Analysis 10: Comparison: Etrasimod 2 mg vs Placebo; Week 48; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 30.00, 95% CI 2-sided [20.97 to 39.03]
Statistical Analysis 11: Comparison: Etrasimod 2 mg vs Placebo; Week 52; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 26.84, 95% CI 2-sided [17.60 to 36.07]

22. Secondary Outcome: Percentage of Participants Achieving 4-week Corticosteroid-free Clinical Remission at Week 52 Among Participants Receiving Corticosteroids at Baseline
Description: Four-week corticosteroid-free clinical remission was defined as an SF subscore = 0 (or = 1 with a ≥ 1-point decrease from Baseline), RB subscore = 0, and ES ≤ 1, and have not received corticosteroids for ≥ 4 weeks in the 40-Week Treatment Period. Each component subscore ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: At Week 52
Population: FAS with actual Baseline MMS 5 to 9. Only participants receiving corticosteroids at study entry and who had not been receiving corticosteroids for ≥ 4 weeks prior to Week 52 were included in this analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 87 | 40
Percentage of participants | 31.0 | 7.5
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 23.05, 95% CI 2-sided [10.20 to 35.90]

23. Secondary Outcome: Percentage of Participants Achieving Clinical Remission at Week 52 Among Participants in Clinical Response at Week 12
Description: Clinical remission and clinical response were based on the MMS which is a composite of 3 assessments: SF, RB and ES. Clinical remission was defined as an SF subscore = 0 (or = 1 with a ≥ 1-point decrease from Baseline), RB subscore = 0, and ES ≤ 1 (excluding friability). Clinical response was defined as a ≥ 2-point and ≥ 30% decrease from Baseline MMS, and a ≥ 1-point decrease from Baseline in RB subscore or an absolute RB subscore ≤ 1. Each component subscore ranged from 0 to 3 and total score range of the MMS was from 0 to 9, with higher scores indicating more severe disease.
Time Frame: At Week 52
Population: FAS with actual Baseline MMS 5 to 9. Only participants in clinical response at Week 12 were included in this analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Etrasimod 2 mg | Placebo
Number analyzed (Participants) | 171 | 46
Percentage of participants | 49.1 | 17.4
Statistical Analysis 1: Comparison: Etrasimod 2 mg vs Placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 31.86, 95% CI 2-sided [18.45 to 45.28]

ADVERSE EVENTS:
Time Frame: Up to 56 weeks (12-Week and 40-Week Treatment Periods plus Follow-up). Treatment-emergent adverse events (TEAEs) were collected from first dose of study treatment up to 30 days following discontinuation of the study treatment.
Description: TEAEs, defined as those adverse events that started or worsened in severity after the first dose of study treatment, are reported for the Safety Population which included all randomized participants who received at least 1 dose of study treatment.
Arm/Group | Etrasimod 2 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/289 | 0/144
Serious Adverse Events (participants affected / at risk) | 20/289 | 9/144
Other Adverse Events (participants affected / at risk) | 204/289 | 77/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etrasimod 2 mg (N=289) | Placebo (N=144)
Colitis ulcerative (Gastrointestinal disorders) | 6 | 3
Mucosal prolapse syndrome (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Peritonitis (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Breast conserving surgery (Surgical and medical procedures) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etrasimod 2 mg (N=289) | Placebo (N=144)
COVID-19 (Infections and infestations) | 19 | 8
Respiratory tract infection viral (Infections and infestations) | 6 | 2
Urinary tract infection (Infections and infestations) | 6 | 3
COVID-19 pneumonia (Infections and infestations) | 4 | 1
Cystitis (Infections and infestations) | 4 | 0
Bronchitis (Infections and infestations) | 3 | 0
Pharyngitis (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4
Anal abscess (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Herpes zoster (Infections and infestations) | 2 | 0
Candida infection (Infections and infestations) | 2 | 1
Hordeolum (Infections and infestations) | 2 | 0
Oral herpes (Infections and infestations) | 2 | 1
Pustule (Infections and infestations) | 2 | 0
Conjunctivitis (Infections and infestations) | 1 | 4
Abscess limb (Infections and infestations) | 1 | 0
Acne pustular (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Helminthic infection (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Pulpitis dental (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Tinea infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Ear infection staphylococcal (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 1
Vulval abscess (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 17 | 10
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Flatulence (Gastrointestinal disorders) | 6 | 0
Abdominal pain (Gastrointestinal disorders) | 11 | 5
Abdominal distension (Gastrointestinal disorders) | 4 | 3
Haemorrhoids (Gastrointestinal disorders) | 7 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 4 | 1
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0
Anal pruritus (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0
Aphthous ulcer (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Abdominal tenderness (Gastrointestinal disorders) | 1 | 1
Proctalgia (Gastrointestinal disorders) | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 2 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Mucosal prolapse syndrome (Gastrointestinal disorders) | 1 | 0
Rectal tenesmus (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Small intestine polyp (Gastrointestinal disorders) | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 3
Blood creatine phosphokinase increased (Investigations) | 5 | 1
Alanine aminotransferase increased (Investigations) | 8 | 2
Gamma-glutamyltransferase increased (Investigations) | 5 | 2
Transaminases increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 3
SARS-CoV-2 test positive (Investigations) | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Serum ferritin decreased (Investigations) | 2 | 0
Blood triglycerides increased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 2 | 1
Blood cholesterol increased (Investigations) | 2 | 0
Weight increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 1 | 1
Blood iron decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 1
C-reactive protein increased (Investigations) | 1 | 0
Blood triglycerides abnormal (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 1
Urine ketone body (Investigations) | 1 | 0
Forced expiratory volume decreased (Investigations) | 1 | 0
Bacterial test positive (Investigations) | 0 | 1
Spirometry abnormal (Investigations) | 1 | 0
FEV1/FVC ratio decreased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 0 | 1
Lung diffusion test decreased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1
Pulmonary arterial pressure decreased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 24 | 7
Dizziness (Nervous system disorders) | 15 | 1
Head discomfort (Nervous system disorders) | 2 | 0
Migraine (Nervous system disorders) | 3 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Asterixis (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Dizziness exertional (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Ankle deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 24 | 14
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 1
Hypocoagulable state (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Pyrexia (General disorders) | 14 | 6
Asthenia (General disorders) | 7 | 2
Fatigue (General disorders) | 5 | 2
Chest discomfort (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 2 | 1
Pain (General disorders) | 2 | 1
Peripheral swelling (General disorders) | 2 | 0
Vaccination site pain (General disorders) | 2 | 0
Discomfort (General disorders) | 1 | 0
Drug intolerance (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 2
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Infusion site reaction (General disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Malaise (General disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Iron deficiency (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Lipomatosis (Metabolism and nutrition disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0
Alopecia scarring (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Ephelides (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura senile (Skin and subcutaneous tissue disorders) | 1 | 0
Xanthelasma (Skin and subcutaneous tissue disorders) | 1 | 0
Papilloedema (Eye disorders) | 2 | 0
Vision blurred (Eye disorders) | 2 | 0
Cataract (Eye disorders) | 3 | 1
Myopia (Eye disorders) | 2 | 0
Amblyopia (Eye disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Astigmatism (Eye disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Eyelid pain (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Eyelid cyst (Eye disorders) | 1 | 0
Macular oedema (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1
Keratitis (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Maculopathy (Eye disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 8 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 2 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Injury corneal (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 1
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 1
Bradycardia (Cardiac disorders) | 4 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Palpitations (Cardiac disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 2
Sleep disorder (Psychiatric disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 1
Cushingoid (Endocrine disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Thyroid cyst (Endocrine disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 1
Primary biliary cholangitis (Hepatobiliary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Micturition frequency decreased (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Penile curvature (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03945188/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/88/NCT03945188/SAP_001.pdf